CLINICAL TRIAL: NCT06311201
Title: Effect of Pilates Exercises on Diastasis Recti Abdominis in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Esam Ghareeb Hasan, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004256
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Diastasis Recti
Keywords: Pilates Exercises; Diastasis Recti Abdominis; Postpartum Women
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal belt (Active Comparator): It consisted of 25 postpartum women who wore abdominal belt for 8 weeks.
  Interventions: Other: Abdominal belt
- Abdominal belt + Pilates exercises (Experimental): It consisted of 25 postpartum women who followed Pilates training program, 3 times/week for 1 hour the session in addition to wearing abdominal belt, for 8 weeks
  Interventions: Other: Abdominal belt; Other: Pilates exercises

INTERVENTIONS:
Other: Abdominal belt — This was used for all women in both groups (A and B) for 8 weeks starting from the 7th days after delivery. The women was asked to wear the abdominal belt throughout the day except when bathing, eating and sleeping. The binder was worn over the skin directly or on a thin layer of clothing. The side of the abdominal binder without the straps was pulled over by the woman's stomach with one hand. The side of the binder with straps was stretched across the stomach and pulled to the center of the abdomen. The straps then was fitted into the buckles. Women were instructed not to wear the binder too tight or too loose as it might irritate the skin and produce difficulty in breathing creating discomfort. They were asked to inspect their skin regularly for any signs of sensitivity.
Other: Pilates exercises — The Pilates exercise program for the study group (B) consisted of a 10-minute warm-up with low-intensity exercises, followed by a 40-minute central part with floor exercises like leg circles, kicks, and stretches. It included the classic "hundred" exercise, performed with proper form. Each exercise had two sets of 10 repetitions. The session ended with a 10-minute cool-down of stretching exercises, supervised by a physical therapist. The program was conducted three times per week, one hour per session, for eight weeks, starting from the 7th day after delivery.
  Arms: Abdominal belt + Pilates exercises

SUMMARY:
The purpose of the study was to investigate the effect of Pilates exercises on diastasis recti abdominis in postpartum women.

DETAILED DESCRIPTION:
Rectus diastasis is relatively common having negative health consequences for women during and after pregnancy (ante-and postnatal periods). Varying estimates of incidence of rectus diastasis have been reported ranging from 66% to 100% during the third trimester of pregnancy, and up to 53% immediately after delivery. Among patients with urogynecological disorders, 52% were found to have a rectus diastasis and 66% had at least one type of pelvic floor dysfunction.

A diastasis can contribute to lower back pain and strain due to other muscles being overworked or compensating for the lack of integrity of abdominals, unstable core, pelvic and back muscles, poor posture, shallow breathing and uterine prolapse. This may result in altered trunk mechanics, impaired pelvic stability and changed posture, which leave the lumbar spine and pelvis more vulnerable to injury.

Facilitation, concentric activation, and stabilization of the abdominal muscles occurred during core stability exercise are used to correct diastasis recti. Pilates has been known to improve the strength and flexibility of muscles, particularly the abdominal muscles, lower back, hip and buttocks i.e. the core musculature thus helping in improving core stability.

Uptill now, there was no previous studies have examined the impact of Pilates training on rectus abdominis diastasis in postpartum women. So, this study will be valuable benefits for medical services organizations and will increase body of knowledge of physical therapists in scientific field.

ELIGIBILITY:
Inclusion Criteria:

1. Postpartum women (7 days after delivery) having diastasis recti (separation between the two recti more than 2.5cm at the level of umbilicus).
2. Multiparous women (2-3) times delivered vaginally with or without episiotomy.
3. Their age ranged from 20 -35 years old.
4. Their BMI was less than 30 kg/cm2.

Exclusion Criteria:

1. Abdominal or back surgery.
2. Abdominal hernia.
3. History of abnormal pregnancy, uterine fibroid or polyhydraminos during pregnancy.
4. Neurological disorders as multiple sclerosis, stroke and spinal lesion.
5. Musculoskeletal diseases such as fractures muscle strains, severe knee osteoarthritis which may affect their physical activity.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Measurement of separation between the two-rectus abdominis muscles above the umbilicus at rest | 8 weeks
  The distance between the recti muscles was measured 4.5 cm above the umbilicus at rest at the beginning and again at the end of the study duration.
Measurement of separation between the two-rectus abdominis muscles above the umbilicus during contraction | 8 weeks
  The distance between the recti muscles was measured 4.5 cm above the umbilicus during contraction at the beginning and again at the end of the study duration.
Measurement of separation between the two-rectus abdominis muscles at level of the umbilicus at rest | 8 weeks
  The distance between the recti muscles was measured at level of the umbilicus at rest at the beginning and again at the end of the study duration.
Measurement of separation between the two-rectus abdominis muscles at level of the umbilicus during contraction | 8 weeks
  The distance between the recti muscles was measured at level of the umbilicus during contraction at the beginning and again at the end of the study duration.
Measurement of separation between the two-rectus abdominis muscles below the umbilicus at rest | 8 weeks
  The distance between the recti muscles was measured 4.5 cm below the umbilicus at rest at the beginning and again at the end of the study duration.
Measurement of separation between the two-rectus abdominis muscles below the umbilicus during contraction | 8 weeks
  The distance between the recti muscles was measured 4.5 cm below the umbilicus during contraction at the beginning and again at the end of the study duration.
Assessment of trunk flexion strength | 8 weeks
  Trunk flexion strength was graded from 0 to 5 using Daniels and Worthingham's procedure before and after the end of the study program. For grades 3-5, the patient curled up through the full range of motion until the scapulae cleared the table. For grade 2, the patient just lifted their head off the table. For grades 0 and 1, the therapist used assisted forward lean or coughing techniques while palpating the rectus abdominis.
Assessment of static trunk flexion endurance | 8 weeks
  It was tested before and after the end of the study program by adopting the most challenging position that was achieved in the strength test, and instructing the participating women to hold that position as long as possible. Standardized verbal encouragement was provided by the assessor, and the holding time was determined using a stopwatch. Three repetitions of the static endurance test were performed with at least 3 minutes of rest between trials; the best (longest holding time) of the three trials was used to represent the participant's endurance. The same position used to evaluate trunk flexion endurance at the initial evaluation was used in subsequent evaluations, even if the woman's strength grade improved between evaluations.

SECONDARY OUTCOMES:
Assessment of functional status | 8 weeks
  All participating women with diastasis recti in both groups (A & B) were asked to fill the Inventory of functional status after childbirth questionnaire before and after the end of the study program. This questionnaire includes five domains and 36 items, that is, infant care (6 items), personal care (8 items), household activities (12 items), social and community activities (6 items), and occupational activities (4 items). The questionnaire was rated on a 4-point Likert scale and the mean score was calculated with one point being the lowest and four points being the highest scores possible. Higher scores indicated better functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Azza BN Kassab, Prof., Study Chair — Cairo University
Locations (1):
- Cairo University, Giza, Egypt